CLINICAL TRIAL: NCT04941885
Title: A Phase II Single-arm Clinical Trial of the Efficacy and Tolerability of Inetetamab Combined With Cyclophosphamide Metronomic Chemotherapy and Aromatase Inhibitor in Metastatic HER2+/HR+ Breast Cancer
Brief Title: Inetetamab Plus Cyclophosphamide Metronomic Chemotherapy Plus Aromatase Inhibitor in Metastatic HER2+/HR+ Breast Cancer
Acronym: Increase
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wang shusen, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-2021
Record Dates: First submitted 2021-06-25; First posted 2021-06-28 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inetetamab Plus Cyclophosphamide Metronomic Chemotherapy Plus AI (Experimental): Each participant receives Inetetamab(8mg/kg iv day 1 followed by 6mg/kg iv day 1, cycled every 21 days) plus cyclophosphamide metronomic chemotherapy(50mg once a day orally) plus aromatase(once a day orally).
  Interventions: Drug: Inetetamab Plus Cyclophosphamide Metronomic Chemotherapy Plus AI

INTERVENTIONS:
Drug: Inetetamab Plus Cyclophosphamide Metronomic Chemotherapy Plus AI — Each participant receives Inetetamab plus cyclophosphamide metronomic chemotherapy plus AI.

SUMMARY:
Antibody-dependent cell-mediated cytotoxicity (ADCC) is one of the important mechanisms for suppressing tumors of Trastuzumab. Pre-clinical data suggest that the ADCC effect of Inetetamab, an anti-HER2 monoclonal antibody with a modified Fc segment, is 1.11 times that of trastuzumab. Previous studies indicated that enhanced ADCC effects can be transformed into clinical benefits. Immune induction through cyclophosphamide metronomic chemotherapy may further enhance the ADCC effect of anti-HER2 monoclonal antibodies. Therefore, we conducted this study to explore the efficacy and the safety of Inetetamab combined with cyclophosphamide metronomic chemotherapy and aromatase inhibitors(AI) in the treatment of metastatic HER2-positive and HR-positive breast cancer patients and to explore the possible mechanisms.

DETAILED DESCRIPTION:
Trastuzumab is a humanized monoclonal antibody, and antibody-dependent cell-mediated cytotoxicity (ADCC) is one of its important mechanisms for suppressing tumors. Pre-clinical data suggest that the ADCC effect of Inetetamab, an anti-HER2 monoclonal antibody with a modified Fc segment, is 1.11 times that of trastuzumab. Previous studies indicated that enhanced ADCC effects can be transformed into clinical benefits, but the absolute benefits are still unsatisfactory. Further improvement of ADCC effects and monoclonal antibody-induced immune responses may improve the clinical benefits. Immune induction through cyclophosphamide metronomic chemotherapy may further enhance the ADCC effect of anti-HER2 monoclonal antibodies. According to previous clinical studies, for HR-positive and HER2-positive metastatic breast cancer patients, metronomic chemotherapy combined with endocrine therapy and anti-HER2 targeted therapy may be one of the treatment options. Therefore, we conducted this study to explore the efficacy and the safety of Inetetamab combined with cyclophosphamide metronomic chemotherapy and aromatase inhibitors(AI) in the treatment of metastatic HER2-positive and HR-positive breast cancer patients, and we further exploring the possible mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form;
2. 18-75 years old;
3. The expected survival period is ≥12 weeks;
4. Eastern Cooperative Oncology Group (ECOG) score [0-2] points;
5. The diagnosis of invasive carcinoma by histology or cytology; Estrogen receptor (ER) positive (defined as >1% nuclear ER staining); HER2 negative (defined as IHC 0 or 1+, or HER2(2+) with HER2 FISH detection no amplification);
6. Inoperable or recurrent/metastatic breast cancer patients with aromatase inhibitor treatment failure;
7. In the state of disease progression before enrollment;
8. Measurable disease according to RECIST version 1.1 or only bone metastasis;
9. Adequate hematological, hepatic and renal function;
10. NYHA class I or II and Left ventricular ejection fraction (LVEF) ≥50%.
11. The diagnosis of invasive carcinoma by histology or cytology: Hormone receptor (HR) positive (defined as >1% nuclear estrogen receptor staining); HER2 positive (defined as IHC 3+, or HER2 FISH detection amplification);
12. In the state of disease progression before enrollment;
13. Have lesions able to and agree to perform tissue biopsy at the time requested in the study;
14. Treatment ≥1 line after recurrence/metastasis, or relapse within 12 months after completing trastuzumab-based adjuvant therapy or during trastuzumab adjuvant therapy;
15. Previously received trastuzumab for anti-HER2 therapy;
16. Measurable disease according to RECIST version 1.1.

Exclusion Criteria:

1. Allergic to the ingredients of Inetetamab, cyclophosphamide or similar drugs;
2. Concomitant diseases/conditions that is not controllable, and any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the patient's participation in this study;
3. Patients who cannot accept drugs orally;
4. Women who are pregnant or breastfeeding or planning to give birth;
5. Patients with currently symptomatic brain or meningeal metastasis;
6. History of other primary malignancy;
7. Resistant to steroidal or nonsteroidal aromatase Inhibitor;
8. Have used Inetetamab;
9. Patients with life-threatening, symptomatic, metastatic visceral disease.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-06-25 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  The proportion of best overall response of either complete or partial response.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | 1 year
  Response and progression will be evaluated using RECIST 1.1. Evaluation will occur every 3 months till progression or termination of the study. CBR is defined as ratio of participants who have stable disease for over 24 weeks.
Progression free survival (PFS) | 1 year
  Time from the date of treatment to the date of tumor progression.
Duration of response (DOR) | 1 year
  Time from the first assessment of the tumor as complete or partial response to the first assessment as PD (Progressive Disease) or death from any cause.
Overall survival (OS) | 3 years
  Time from the date of treatment to the date of death.
Number of Participants with Adverse Events | 1 year
  Number of participants with adverse events related to the treatment.
The quality of life | 1 year
  Using Functional Assessment of Cancer therapy -Breast (FACT-B) scale. The minimum and maximum values are 0 and 144, respectively. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Shusen Wang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No